CLINICAL TRIAL: NCT07342595
Title: Clinical Performance of an Intraoral Scanner With Integrated Caries Detection
Brief Title: Evaluation of Radiation-Free Caries Detection Integrated Into Intraoral Scanners Compared With Conventional Diagnostic Methods
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Mehl (Other)
Responsible Party: Sponsor-Investigator, Albert Mehl, Prof. Dr. Dr., University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-01988
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Caries Assessment; Caries; Dentin; Caries; Initial
Keywords: Caries detection; near-infrared light; clinical performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- intraoral scan (Other)
  Interventions: Diagnostic Test: intraoral scan with integrated caries detection tool

INTERVENTIONS:
Diagnostic Test: intraoral scan with integrated caries detection tool — The intervention in this study is the addition of a non-invasive intraoral scan of the tooth scheduled for extraction and its adjacent teeth using the iTero Lumina device. This scan is CE-certified, performed according to the manufacturer's instructions, takes approximately 5 minutes, involves no radiation, and does not change the standard dental treatment. All other procedures, including visual examination, radiographs, and tooth extraction, are part of routine care and are not affected by the study.

SUMMARY:
The goal of this study is to evaluate if an intraoral scanning device with an integrated radiation-free caries detection tool (near-infrared light) can detect early tooth decay.

The main questions it aims to answer are:

Can the tool find tooth decay as accurately as traditional visual and X-ray examinations? How reliable is the tool when used by different dentists?

Participants will:

* Have one tooth scheduled for extraction. This tooth and its adjacent teeth need to be examined before the extraction by using the intraoral scanner with the caries detection tool, which takes about 5 extra minutes. Those results will be compared to the standard dental examination, including visual inspection and X-rays.
* Allow investigators to check the extracted tooth and the neighboring teeth directly after extraction to see if any carious lesion is visible.

This study does not involve any drugs or invasive procedures beyond the planned tooth extraction, and participants will not be exposed to extra radiation. The results will help dentists detect tooth decay, which may allow less invasive treatments and better prevention.

ELIGIBILITY:
Inclusion Criteria:

* All genders, minimum age for participation is 18 years
* Presence of a tooth, that is already scheduled for extraction (indication for extraction diagnosed during the normal clinical service independently of this study by a qualified dentist)
* Availability of a radiograph (X-ray) showing the tooth to be extracted along with adjacent teeth
* Signed informed consent after a comprehensive explanation of the study is available

Exclusion Criteria:

* participants under the age of 18
* Addicts or participants with impaired cognitive abilities that do not allow the participant to assess the scope of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Performance of the caries detection tool, integrated in intraoral scanning system in terms of sensitivity, specificity and reliability. | From the enrollment at four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Mehl, Prof. Dr. Dr., Principal Investigator — University of Zurich, Center for Dental Medicine
Locations (1):
- University of Zurich - Center for Dental Medicine, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
The ethics application, which has already been approved, contains clear provisions on data protection. There is no provision for data to be passed on; accordingly, the investigators must protect all personal data and may not pass it on to third parties.